CLINICAL TRIAL: NCT00005626
Title: Phase II Trial With Correlative Laboratory Studies of Single Agent Irinotecan (Camptosar CPT-11) in Newly Diagnosed and Relapsed Indolent Lymphoproliferative Malignancies
Brief Title: Phase II Trial With Correlative Laboratory Studies of Single Agent Irinotecan (Camptosar CPT-11)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Upjohn (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11586; NCI-G00-1764 (Other: NCI)
Record Dates: First submitted 2000-05-02; First posted 2004-08-10 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Leukemia; Lymphoma
Keywords: stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; prolymphocytic leukemia; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irinotecan Treatment (Experimental): Patients receive irinotecan IV over 90 minutes on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for 2-6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed for survival.
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — Irinotecan as outlined in treatment arm
  Other Names: irinotecan hydrochloride; Camptosar CPT-11

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients who have newly diagnosed or relapsed non-Hodgkin's lymphoma or leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete and partial response rates in patients with newly diagnosed or relapsed indolent non-Hodgkin's lymphoma, high risk chronic lymphocytic leukemia, or prolymphocytic leukemia treated with irinotecan. II. Determine the toxicity of this regimen in these patients. III. Correlate the level of DNA topoisomerase I mRNA and protein, as well as SN-38 induced topoisomerase I-DNA complex formation, with the clinical response and toxicity in these patients. IV. Determine if a down regulation of topoisomerase I or altered subcellular distribution of this enzyme is involved in the drug resistance to irinotecan.

OUTLINE: Patients receive irinotecan IV over 90 minutes on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for 2-6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 17-40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven newly diagnosed or relapsed non-Hodgkin's lymphoma (NHL) of 1 of the following types: Low grade (diffuse small lymphocytic/marginal zone, grade I follicular small cleaved cell, or grade II follicular mixed cell) OR Mantle cell OR Histologically proven newly diagnosed or relapsed stage III or IV chronic lymphocytic leukemia (CLL) or prolymphocytic leukemia (PLL) At least 1 measurable disease parameter Enlarged spleen extending at least 2 cm below the costal margin constitutes measurable disease provided that no explanation other than lymphomatous involvement is likely Enlarged liver extending at least 5 cm below the costal margin constitutes measurable disease Not allowable as sole indication for therapy: Isolated splenomegaly OR Isolated hepatomegaly No central nervous system (CNS) metastases or carcinomatous meningitis A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Eastern Cooperative Oncology Group (ECOG) 0-2 Life expectancy: At least 12 weeks Hematopoietic: NHL: Granulocyte count greater than 1,500/mm^3 Hemoglobin at least 9.0 g/dL Platelet count greater than 100,000/mm^3 CLL or PLL: Granulocyte count greater than 500/mm^3 Hemoglobin greater than 7.0 g/dL Platelet count greater than 50,000/mm^3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN if liver tumor present) No Gilbert's disease Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 60 mL/min Calcium less than 12.0 mg/dL (corrected) Cardiovascular: No myocardial infarction or atrial fibrillation within the past 6 months No congestive heart failure requiring therapy Other: No active or uncontrolled infection HIV negative No psychiatric disorder that would preclude informed consent or compliance No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No history of seizures No uncontrolled diabetes mellitus, defined as random blood glucose at least 200 mg/dL No other severe concurrent disease that would increase risk

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior irinotecan or any other topoisomerase I inhibitor (e.g., topotecan) Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No concurrent phenytoin, phenobarbital, or other antiepileptic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 1998-02; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 5 years
  Objective Response Rate according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Determine the complete and partial response rates in patients with newly diagnosed or relapsed indolent non-Hodgkin's lymphoma, high risk chronic lymphocytic leukemia, or prolymphocytic leukemia treated with irinotecan.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 5 years
  Review of adverse events utilizing Common Toxicity Criteria (CTC) V3.

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Goldstein, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States